CLINICAL TRIAL: NCT06435572
Title: Effect of Open and Closed Suction Systems on Newborn's Pain and Vital Signs in Neonatal Intensive Care
Brief Title: Comparison of Open and Closed Aspiration in Newborns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Aslı Alaca, MSc, Izmir Katip Celebi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: aslialaca
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Newborn
Keywords: Closed system suctioning; Open system suctioning; Pain; Neonatal intensive care; Newborn; Suction
MeSH Terms: conditions — Pain | interventions — Suction

STUDY DESIGN:
Intervention Model Description: Each patient will be considered as both an experimental and a control group.Two different aspiration methods will be applied in line with the patient's aspiration needs, and the effect of the methods will be evaluated on the same patient. In the study, open aspiration applied to the patient will be evaluated as control, and closed aspiration will be considered as the experimental group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental and A control group (Experimental): Each patient will be evaluated as both the experimental and control group. In line with the patient's aspiration needs, two different suction methods will be applied and the effects of the methods will be evaluated on the same patient. In the study, open suction applied to the patient will be considered as the control group, and closed suction will be considered as the experimental group. The first suction of the same patient during the day will be performed as open suction, and the second suction will be performed as closed suction. Pain and physiological parameters will be evaluated before, during and 30 minutes after each sucking session.
  Interventions: Other: Suction

INTERVENTIONS:
Other: Suction — Each patient will be evaluated as both the experimental and control group. In the study, open suction applied to the patient will be evaluated as control, and closed suction will be considered as the experimental group. The first suction of the same patient during the day will be done as open suction, and the second suction will be done as closed suction.
  Other Names: open suction; closed suction

SUMMARY:
Endotracheal aspiration is a necessary procedure performed by nurses in neonatal intensive care units to increase oxygenation and remove secretions from the airways. It is one of the painful procedures that most frequently causes stress in intubated newborns.

DETAILED DESCRIPTION:
The aim of this study is to examine the effect of open and closed system suction, which is one of the invasive procedures frequently applied in neonatal intensive care, on the baby's pain and vital signs. There is a need for innovative, evidence-based practices to be implemented by nurses in clinics to minimize complications related to endotracheal suction.

ELIGIBILITY:
Inclusion Criteria:

* Newborns monitored with mechanical ventilation
* Newborn who need suctioning,
* Newborn who did not undergo painful procedures one hour before aspiration.
* Hemodynamically stable newborn;

Exclusion Criteria:

* Newborn with any facial/skull deformities
* Newborn with chromosomal/genetic abnormalities

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-21 (Estimated); Primary Completion 2025-06-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Pain score | Pain will be evaluated before, during and 30 minutes after each suction procedure.
  differences in pain between open and closed suctioning systems
Oxygen saturation | Oxygen saturation will be evaluated before, during and 30 minutes after each suction procedure
  differences in oxygen saturation between open and closed suctioning systems
Heart rate | Heart rate will be evaluated before, during and 30 minutes after each aspiration procedure
  differences in heart rate between open and closed suctioning systems

CONTACTS AND LOCATIONS:
Locations (1):
- Aslı Alaca, Buca, İ̇zmi̇r- Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No